CLINICAL TRIAL: NCT01250665
Title: Cohort Study Comparing Corpus Callosum Atrophy as a Marker of Later Development of Cognitive Impairment in Patients With Early and Remitting Relapsing Multiple Sclerosis
Brief Title: Study Comparing Corpus Callosum Atrophy as a Marker of Later Development of Cognitive Impairment in Patients With Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cantonal Hospital of St. Gallen (Other)
Collaborators: Bayer (Industry)
Responsible Party: Murat Yildiz, Cantonal Hospital Saint Gallen
Other Study IDs: CogImp01
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Multiple Sclerosis; Cognitive Impairment
Keywords: multiple sclerosis; cognitive impairment; interferon-beta 1b; corpus callosum index
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- clinically isolated syndrome: In this study the term clinically isolated syndrome (CIS) is defined according to the Task Force on Differential Diagnosis in MS, as a monophasic presentation of neurological symptoms with suspected underlying inflammatory demyelinating disease (Miller 2008).
- remitting, relapsing MS: remitting relapsing MS according to the criteria by Poser (Poser 1983) or McDonald (McDonald 2001)

SUMMARY:
This study is a cross sectional study of patients diagnosed with clinically isolated syndrome (CIS) and RRMS, who will undergo a series of tests to assess cognitive impairment, fatigue severity and depressive symptoms. Cognitive impairment will be assessed with Multiple Sclerosis Inventory Cognition (MUSIC) and symbol digit modalities test (SDMT), fatigue severity will be measured with the Fatigue Scale for Motor and Cognitive Functions (FSMC) and depressive symptoms with the Beck Depression Inventory (BDI). All tests mentioned above are validated for MS patients. In the second step we will use our large longitudinal database of serial MRI examinations from which a linear measurement of CCI will be retrospectively calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 55 years at presentation
* Diagnosis of relapsing-remitting MS according to revised McDonald criteria 2005, clinically isolated syndrome suggestive of MS
* Patients treated with interferon-beta 1b
* Untreated patients
* EDSS under 5.5

Exclusion Criteria:

* Brain pathology other than MS
* Known history of head trauma
* Pure spinal manifestation of demyelization
* Neuromyelitis optica
* Primary and secondary progressive MS
* Benzodiazepine intake within the last three months
* Relapse within the last three months
* Steroid intake within the last three months
* History of severe depressive disorder and/or suicidality, seizure, drug or alcohol abuse
* No informed consent
* Insufficient knowledge of German

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: MS-Patients will be recruited in the outpatient clinic of the neurology department of the cantonal hospital of Saint Gallen, responsible for treatment of MS patients of Northeast Switzerland.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Multiple Sclerosis Inventory Cognition (MUSIC)
  MUSIC is a cognitive screening instrument. It assesses the cognitive core deficit in MS (mental flexibility, attention, information processing speed, memory and inhibitory control) and includes 3 items derived from a factorial analysis to examine cognitive, motor and psychosocial fatigue, respectively.
Annual Corpus Callosum Index decrease
  Corpus callosum index (CCI) is an easy to use MRI marker for estimating brain atrophy in patients with MS. Demonstrated correlation of CCI and atrophy has been measured with brain parenchymal fraction.

SECONDARY OUTCOMES:
Corpus callosum Index at baseline
  The CCI at baseline will be measured from MRI findings acquired at diagnosis of clinically isolated syndrome.
Time to clinically definite MS
  This is the time in months then patients diagnosed with CIS go on to develop clinically definite MS (CDMS). CDMS will be diagnosed if patients fulfill the criteria for remitting relapsing MS according to Poser (Poser 1983) or McDonald (McDonald 2001).
The Symbol Digit Modalities Test (SDMT)
  SDMT is an easily administered brief cognitive performance tests. This test emphasizes working memory and speed processing.
Ratio treatment duration to disease duration
  The ratio of duration of treatment (DT) to duration of disease (DD): DT/DD. Duration of treatment is the cumulative time of treatment with interferon-beta 1b. Duration of disease starts from the first presentation of MS symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Murat Yildiz, MD, Principal Investigator — Cantonal Hospital Saint Gallen
Locations (1):
- Cantonal Hospital of Saint Gallen, Sankt Gallen, Switzerland

REFERENCES:
- [Derived] Yildiz M, Tettenborn B, Radue EW, Bendfeldt K, Borgwardt S. Association of cognitive impairment and lesion volumes in multiple sclerosis--a MRI study. Clin Neurol Neurosurg. 2014 Dec;127:54-8. doi: 10.1016/j.clineuro.2014.09.019. Epub 2014 Oct 14. PMID 25459243